CLINICAL TRIAL: NCT05996289
Title: Inter-observer Variability in the Segmentation of Prostate Tumour Lesions Using Multiparametric MRI
Brief Title: Inter-observer Variability in the Segmentation of Prostate Tumour Lesions Using Multiparametric MRI (VARIOP)
Acronym: VARIOP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC23.0145 - VARIOP
Record Dates: First submitted 2023-08-01; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer
Keywords: radiotherapy; MRI; segmentation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Following the major technological and scientific advances in external radiotherapy in recent decades, thanks to the use of three-dimensional conformal techniques combined with intensity modulation, image-guided radiotherapy has enabled radiotherapists to increase doses without increasing sequelae and complications, giving rise to the term "dose escalation".

Following multiple dose-escalation clinical trials showing better biological control of PSA, the results of the latest phase 3 FLAME trial incorporated the notion of intraprostatic boost in relation to the primary prostate lesion, considered to be the preferred site of neoplastic recurrence in prostate cancer.

This leads to the first question, which concerns the identification of the dominant lesion and its precise delimitation. This last point is subject to variation between operators. A retrospective cohort from the Finistère region will therefore be used to develop a number of study points relating to :

inter-operator contour variability

* Factors influencing contour
* Impact of contour variability on dosimetry
* Automatic segmentation

DETAILED DESCRIPTION:
Following the major technological and scientific advances in external radiotherapy in recent decades, thanks to the use of three-dimensional conformal techniques combined with intensity modulation, image-guided radiotherapy has enabled radiotherapists to increase doses without increasing sequelae and complications, giving rise to the term "dose escalation".

Following multiple dose-escalation clinical trials showing better biological control of PSA, the results of the latest phase 3 FLAME trial incorporated the notion of intraprostatic boost in relation to the primary prostate lesion, considered to be the preferred site of neoplastic recurrence in prostate cancer.

One of the issues raised by such a study is the methodology used to contour the tumour lesion, an issue which concerns the whole field of radiotherapy. The reference imaging technique for diagnosing prostate cancer, and more specifically the dominant tumour lesion, is multiparametric Magnetic Resonance Imaging. This leads to the first question, which concerns the identification of the dominant lesion and its precise delimitation. This last point is subject to variation between operators. A retrospective cohort from the Finistère region will therefore be used to develop a number of study points relating to :

inter-operator contour variability

* Factors influencing contour
* Impact of contour variability on dosimetry
* Automatic segmentation

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically proven localized prostatic neoplasia on trans-rectal biopsies.
* Multiparametric prostate MRI performed prior to prostate biopsies.
* No opposition expressed
* Patient affiliated to a social security scheme

Exclusion Criteria:

* History of surgery, prostatic irradiation or hormonal treatment prior to diagnosis.
* History of prostate cancer
* No identifiable target lesion on mpMRI (<PIRADS 3)
* Opposition formulated
* Patient under legal protection (guardianship, curatorship, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient treated or being treated for prostatic adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Inter-observer variability | through study completion, an average of 6 months
  The main criterion for judging inter-observer variability is the spatial overlap of contours on mpMRI, represented by the DICE similarity coefficient, which ranges from 0 to 1, where 1 represents zero variability between contours of the same lesion.

SECONDARY OUTCOMES:
Clinical factors influencing inter-observer variability. | through study completion, an average of 6 months
  Subgroup analysis of radio-clinical-histological factors likely to influence inter-observer variability.
Assessing inter-sequence reproducibility | through study completion, an average of 6 months
  Assessing inter-sequence reproducibility
Dosimetric impact of Inter-observer variability | through study completion, an average of 6 months
  The influence of variability on dosimetry in IMRT/VMAT conformal radiotherapy.

OTHER OUTCOMES:
Automatic segmentation of prostatic tumors | through study completion, an average of 6 months
  Contour variability using a deep-learning automated segmentation technique, with and without implementation of factors identified as impacting contour in manual technique.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Bourbonne, MD, PhD, Principal Investigator — Radiation Oncology Department, Brest University Hospital
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement